CLINICAL TRIAL: NCT01008774
Title: A Comparison of Different Scalp Cooling Systems for the Prevention of Chemotherapy Induced Alopecia
Brief Title: START: Swiss Taxotere Alopecia Prevention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DOCET_L_04449
Record Dates: First submitted 2009-10-01; First posted 2009-11-06 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Neoplasms; Alopecia
MeSH Terms: conditions — Neoplasms; Alopecia

ARMS (3):
- A (Experimental)
  Interventions: Device: Paxman Cooling Machine
- B (Active Comparator)
  Interventions: Device: Cold Caps
- C (No Intervention)

INTERVENTIONS:
Device: Paxman Cooling Machine — Scalp cooling procedures
  Arms: A
Device: Cold Caps — Scalp cooling procedures
  Arms: B

SUMMARY:
Primary objective:

* Rate of complete chemotherapy induced alopecia (WHO grade III or IV, physician grading)

Secondary objective:

* Compliance to scalp cooling procedure
* Received number of cycles of chemotherapy in each subgroup
* Patient perception of scalp cooling procedure
* Side effects of scalp cooling systems

ELIGIBILITY:
Inclusion Criteria:

* Any solid tumor malignancy receiving docetaxel (Taxotere®) 1st line chemotherapy treatment with the exception of regimen containing concomitant anthracycline treatment; sequential anthracycline/docetaxel treatment is permitted.
* Performance Status ECOG <= 2
* Absence of alopecia at inclusion

Exclusion Criteria:

* Chemotherapy regimen including concomitant anthracycline treatment
* Raynaud's disease or phenomenon
* Cold agglutinin disease
* Cryoglobulinemia
* Cryofibrinogenemia
* Scalp metastasis
* Pregnancy or Lactation
* Preexisting alopecia of any grade; notably androgenetic alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Grade III or IV alopecia according to the WHO criteria | D1 of each cycle and D+21 after last cycle of chemotherapy

SECONDARY OUTCOMES:
Compliance to scalp cooling procedure | D1 of each cycle and D+21 after last cycle of chemotherapy
Side effects of scalp cooling systems | D1 of each cycle and D+21 after last cycle of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- [Derived] Betticher DC, Delmore G, Breitenstein U, Anchisi S, Zimmerli-Schwab B, Muller A, von Moos R, Hugli-Dayer AM, Schefer H, Bodenmann S, Buhler V, Trueb RR. Efficacy and tolerability of two scalp cooling systems for the prevention of alopecia associated with docetaxel treatment. Support Care Cancer. 2013 Sep;21(9):2565-73. doi: 10.1007/s00520-013-1804-9. Epub 2013 May 2. PMID 23636645